CLINICAL TRIAL: NCT06945549
Title: Evaluation of Intestinal Lesions and Disease Activity in Inflammatory Bowel Disease Based on 18F-FAPI PET Imaging
Acronym: IBD，18F-FAPI
Status: Recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025137
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Disease (IBD); Disease Activity; FAPI
Keywords: Inflammatory bowel disease; 18F-FAPI PET; disease activity
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBD patient group: Patients diagnosed with IBD according to clinical, imaging, endoscopic, and histopathological criteria.
  Interventions: Diagnostic Test: 18F-FAPI PET Imaging

INTERVENTIONS:
Diagnostic Test: 18F-FAPI PET Imaging — The ROI of the target lesions was delineated based on 18F-FAPI PET Imaging, and the lesions were divided on the cross section to obtain the lesions SUVmax, SUVmean, SUVpeak, FAPI metabolic volume (FAV), MTV, TBR, and TLG.

SUMMARY:
The goal of this observational study is to evaluate the role and effect of 18F-FAPI PET imaging in the identification of intestinal lesions and the assessment of disease activity in inflammatory bowel disease. The main question it aims to answer is:

Can 18F-FAPI PET imaging effectively identify intestinal lesions in inflammatory bowel disease and accurately assess disease activity? Colonoscopy, enhanced abdominal CT, and 18F-FAPI intestinal imaging were completed within 1 week, and major adverse outcomes (MAO) were followed up 12 months after enrollment.

Last updated on March 25, 2025

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with IBD according to clinical, imaging, endoscopic, and histopathological criteria;
* Patients ≥18 years old;
* 18F-FAPI PET/CT intestinal imaging, conventional endoscopic and enhanced CT were performed within 1 week;
* Intestinal segment matching was evaluated by endoscopy and imaging;
* Patients voluntarily participate and sign informed consent.

Exclusion Criteria:

* Pregnant or lactating patients;
* Imaging images are of poor quality and cannot be used for diagnosis and evaluation;
* Patients with contraindications for endoscopic or CT examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IBD according to clinical, imaging, endoscopic, and histopathological criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of 18F-FAPI PET imaging and enhanced CT in the identification of intestinal lesions in IBD was compared and evaluated | 2025.4-2027.12
  The sensitivity and specificity of PET/ CT and enhanced CT to detect endoscopic lesions were calculated and compared by receiver operating characteristic (ROC) curves.
Association of 18F-FAPI imaging with endoscopic disease activity | 2025.4-2027.12
  Spearman test was used to evaluate the correlation between overall FAPI PET/CT score and IBD endoscopic range of motion (modified Mayo endoscopic score, UCEIS).
The difference of FAPI SUVmax among different endoscopic MES evaluation groups | 2025.4-2027.12
  Taking into account multiple intestinal segments in each patient, mixed model ANOVA and Bonferroni-adjusted postmortem tests were performed to compare the differences in SUVmax between different MES rating groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Army Medical Center of PLA, Daping Hospital, Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luo Y, Pan Q, Xu H, Zhang R, Li J, Li F. Active uptake of 68Ga-FAPI in Crohn's disease but not in ulcerative colitis. Eur J Nucl Med Mol Imaging. 2021 May;48(5):1682-1683. doi: 10.1007/s00259-020-05129-7. Epub 2020 Nov 27. No abstract available. PMID 33247327
- [Background] Chen L, Zhong X, Li L, Li X, Liu Y, Guo C, Chen Y, Huang Z. [68Ga]Ga-FAPI-04 PET/CT on assessing Crohn's disease intestinal lesions. Eur J Nucl Med Mol Imaging. 2023 Apr;50(5):1360-1370. doi: 10.1007/s00259-023-06107-5. Epub 2023 Jan 12. PMID 36631715
- [Background] Luo Y, Pan Q, Yang H, Peng L, Zhang W, Li F. Fibroblast Activation Protein-Targeted PET/CT with 68Ga-FAPI for Imaging IgG4-Related Disease: Comparison to 18F-FDG PET/CT. J Nucl Med. 2021 Feb;62(2):266-271. doi: 10.2967/jnumed.120.244723. Epub 2020 Jun 8. PMID 32513902
- [Background] Diekmann J, Koenig T, Thackeray JT, Derlin T, Czerner C, Neuser J, Ross TL, Schafer A, Tillmanns J, Bauersachs J, Bengel FM. Cardiac Fibroblast Activation in Patients Early After Acute Myocardial Infarction: Integration with MR Tissue Characterization and Subsequent Functional Outcome. J Nucl Med. 2022 Sep;63(9):1415-1423. doi: 10.2967/jnumed.121.263555. Epub 2022 Feb 24. PMID 35210301
- [Background] Pang Y, Zhao L, Luo Z, Hao B, Wu H, Lin Q, Sun L, Chen H. Comparison of 68Ga-FAPI and 18F-FDG Uptake in Gastric, Duodenal, and Colorectal Cancers. Radiology. 2021 Feb;298(2):393-402. doi: 10.1148/radiol.2020203275. Epub 2020 Dec 1. PMID 33258746
- [Background] Jacobson FL, Van den Abbeele AD. Importance of 68Ga-FAPI PET/CT for Detection of Cancer. Radiology. 2022 Apr;303(1):200-201. doi: 10.1148/radiol.212884. Epub 2022 Jan 4. No abstract available. PMID 34981981
- [Background] Scharl M, Huber N, Lang S, Furst A, Jehle E, Rogler G. Hallmarks of epithelial to mesenchymal transition are detectable in Crohn's disease associated intestinal fibrosis. Clin Transl Med. 2015 Feb 7;4:1. doi: 10.1186/s40169-015-0046-5. eCollection 2015. PMID 25852817
- [Background] Lovisa S, Genovese G, Danese S. Role of Epithelial-to-Mesenchymal Transition in Inflammatory Bowel Disease. J Crohns Colitis. 2019 Apr 26;13(5):659-668. doi: 10.1093/ecco-jcc/jjy201. PMID 30520951
- [Background] Gordon IO, Bettenworth D, Bokemeyer A, Srivastava A, Rosty C, de Hertogh G, Robert ME, Valasek MA, Mao R, Li J, Harpaz N, Borralho P, Pai RK, Odze R, Feakins R, Parker CE, Guizzetti L, Nguyen T, Shackelton LM, Sandborn WJ, Jairath V, Baker M, Bruining D, Fletcher JG, Feagan BG, Pai RK, Rieder F; Stenosis Therapy and Anti-Fibrotic Research (STAR) Consortium. International consensus to standardise histopathological scoring for small bowel strictures in Crohn's disease. Gut. 2022 Mar;71(3):479-486. doi: 10.1136/gutjnl-2021-324374. Epub 2021 May 5. PMID 33952604
- [Background] Wang J, Lin S, Brown JM, van Wagoner D, Fiocchi C, Rieder F. Novel mechanisms and clinical trial endpoints in intestinal fibrosis. Immunol Rev. 2021 Jul;302(1):211-227. doi: 10.1111/imr.12974. Epub 2021 May 16. PMID 33993489
- [Background] Schmoyer CJ, Saidman J, Bohl JL, Bierly CL, Kuemmerle JF, Bickston SJ. The Pathogenesis and Clinical Management of Stricturing Crohn Disease. Inflamm Bowel Dis. 2021 Oct 20;27(11):1839-1852. doi: 10.1093/ibd/izab038. PMID 33693860
- [Background] Agrawal M, Spencer EA, Colombel JF, Ungaro RC. Approach to the Management of Recently Diagnosed Inflammatory Bowel Disease Patients: A User's Guide for Adult and Pediatric Gastroenterologists. Gastroenterology. 2021 Jul;161(1):47-65. doi: 10.1053/j.gastro.2021.04.063. Epub 2021 Apr 30. PMID 33940007
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/